CLINICAL TRIAL: NCT02282267
Title: Blood Detection of EGFR Mutation For Iressa Treatment
Acronym: Benefit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jie Wang, Chief of thoracic cancer department, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJCHDTC002
Record Dates: First submitted 2014-10-31; First posted 2014-11-04 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Lung Adenocarcinoma
Keywords: Epidermal growth factor receptor; Droplet digital PCR
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Gefitinib

STUDY DESIGN:
Intervention Model Description: Iressa treatment oral daily
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gefitinib (Experimental): Patients with EGFR mutation in plasma detected by droplet digital PCR could receive Gefitinib 250mg every day until disease progression.
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — Iressa 250mg oral daily
  Other Names: Iressa

SUMMARY:
This study was proposed to validate the efficacy of gefitinib as first-line therapy in advanced lung adenocarcinoma with EGFR mutation determined by plasma cf-DNA.

DETAILED DESCRIPTION:
Patients without enough tissue for EGFR mutation detection can also have opportunity to use EGFR-TKI as first line therapy. Meanwhile, this study was also proposed to explore the best intervention time of anti-resistant drugs (such as AZD 9291, a T790M inhibitor) through the quantitative and dynamic analysis of EGFR sensitive and resistant mutation in plasma cf-DNA during EGFR-TKI treatment process.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Male or female patients aged ranging from 18 to 75 years old.
* Histological confirmation of lung adenocarcinoma. Attention: the paraffin embedded cytological samples extracted from pleural effusion are acceptable. Adeno-squamous carcinoma is not allowed to enroll. Sputum cytology alone cannot be acceptable. Bronchoalveolar lavage and fine needle aspiration cytology specimens for lesions also cannot acceptable.
* Metastatic lung adenocarcinoma (stage Ⅳ, IASLC, 2009).
* EGFR sensitive mutation (including exon 19 del and/or exon 21 L858R) in plasma cf-DNA by ddPCR.
* Chemotherapy, immunotherapy and other systemic anti-cancer treatment (such as EGFR inhibitor including other EGFR tyrosine kinase inhibitor and EGFR antibody, and anti-vascular therapy including vascular epithelial growth factor receptor inhibitor and Endostar) naïve. Radical surgery and radiotherapy must be completed at least 6 months before start of study treatment. Adjuvant chemotherapy is allowed and must be finished at least 6months before start of study drug. Palliative radiotherapy must be completed at least 2 weeks before start of study treatment with no persistent radiation toxicity.
* At least one lesion, not previously irradiated, that can be accurately measured at baseline as 10mm in the longest diameter (lymph nodes must have short axis more than 15mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements.
* WHO Performance Status 0, 1 or 2.
* Criteria for laboratory examinations:

Blood white cell count≥3.0*109/L, Neutrophile cell count ≥1.5*109/L Platelet count ≥100*109/L Total bilirubin (TB) ≤ 1.5 times upper limit of normal Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2 times upper limit of normal; for subjects with hepatic metastasis, AST, ALT≤ 5 times upper limit of normal Creatinine clearance≥50ml/min

Exclusion Criteria:

* Known severe allergic to gefitinib or any excipient of the product.
* Considered to require radiotherapy to the lung at the time of study entry or in the near future.
* Newly diagnosed symptomatic central nervous system (CNS) metastasis or spinal cord compression unless treated with surgery and/or radiation and stable without steroid for at least 2 weeks.
* Uncontrolled massive pleural or pericardial effusion.
* Past medical history of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis which required steroid treatment or any evidence of clinically active interstitial lung disease.
* The presence of idiopathic pulmonary fibrosis in baseline CT scans.
* Combined use of phenytoin, rifampin, carbamazepine, pentobarbital or St. John's wort.
* Any obvious ocular anomalies, especially severe dry eye syndrome, keratoconjunctivitis sicca, serious exposure keratitis or other potentially increased epithelial lesions.
* As judged by the investigator, any evidence of severe of uncontrolled systemic disease (e.g. active infection, uncontrolled hypertension unstable angina, congestive hear failure, liver, kidney or metabolic diseases).
* Could not accept oral administration, need intravenous nutrition, previous operation that affect absorption or active peptic ulcer.
* Pregnant or lactating women.
* Prior administration of other study drug or drug without approval within 30 days before the first day of study drug administration.
* Other co-existing malignancies on malignancies diagnosed within the last 5 years, with the exception of basal cell carcinoma or cervical cancer in situ or completely resected intra-mucosal gastric cancer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
objective response rate of gefitinib | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: jie wang, doctor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang Z, Cheng Y, An T, Gao H, Wang K, Zhou Q, Hu Y, Song Y, Ding C, Peng F, Liang L, Hu Y, Huang C, Zhou C, Shi Y, Zhang L, Ye X, Zhang M, Chuai S, Zhu G, Hu J, Wu YL, Wang J. Detection of EGFR mutations in plasma circulating tumour DNA as a selection criterion for first-line gefitinib treatment in patients with advanced lung adenocarcinoma (BENEFIT): a phase 2, single-arm, multicentre clinical trial. Lancet Respir Med. 2018 Sep;6(9):681-690. doi: 10.1016/S2213-2600(18)30264-9. Epub 2018 Jul 17. PMID 30017884